CLINICAL TRIAL: NCT06357364
Title: Neural Changes Following Cognitive Behavior Therapy (CBT) for Procrastination: An fMRI and EEG Randomized Controlled Trial of Two CBT Protocols
Brief Title: Neural Changes Following Cognitive Behavior Therapy for Procrastination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nencki Institute of Experimental Biology of the Polish Academy of Sciences (Other Government)
Collaborators: SWPS University of Social Sciences and Humanities (Other); Institute of Psychology, Polish Academy of Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT_Procrastination_Neuro
Record Dates: First submitted 2024-03-18; First posted 2024-04-10 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Procrastination

STUDY DESIGN:
Who Masked: Participant
Masking Description: A researcher not having direct contact with participants will create a script generating random sequence using a computer random sequence generator (Matlab). Randomization will take place at an individual level, stratified by age, gender and procrastination severity (block randomization). Participants will be randomized into three groups with an allocation ratio of 1:1:1.
  Pairs of experienced psychotherapists trained in one of the therapy protocols will deliver the interventions in an online group setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy with Techniques of Starting on Time and Planning Realistically (Experimental): 5 session (one session a week) online group therapy including psychoeducation and cognitive modules (what is procrastination, role of rewards, work environment, identification of dysfunctional automatic thoughts, cognitive restructuring, relapse prevention) and a behavioral module: realistic planning, timely beginning.
  Interventions: Behavioral: Psychoeducation and cognitive modules; Behavioral: Behavioral module: Starting on Time and Planning Realistically
- Cognitive Behavioral Therapy with Technique of Working Time Restriction (Experimental): 5 session (one session a week) online group therapy including psychoeducation and cognitive modules (what is procrastination, role of rewards, work environment, identification of dysfunctional automatic thoughts, cognitive restructuring, relapse prevention) and a behavioral module: working time restriction.
  Interventions: Behavioral: Psychoeducation and cognitive modules; Behavioral: Behavioral module: Working Time Restriction
- Wait-list control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Psychoeducation and cognitive modules — Psychoeducation and cognitive modules: what is procrastination, role of rewards, work environment, belief identification, cognitive restructuring, relapse prevention.
  Arms: Cognitive Behavioral Therapy with Technique of Working Time Restriction; Cognitive Behavioral Therapy with Techniques of Starting on Time and Planning Realistically
Behavioral: Behavioral module: Starting on Time and Planning Realistically — Learning of realistic planning, and timely starting of work.
  Arms: Cognitive Behavioral Therapy with Techniques of Starting on Time and Planning Realistically
Behavioral: Behavioral module: Working Time Restriction — Restriction of allowed time for work, and gradual increase of allowed time, if previous time windows where effectively used.
  Arms: Cognitive Behavioral Therapy with Technique of Working Time Restriction

SUMMARY:
The aim of this study is to compare the efficacy of and the neural changes following two cognitive behavior therapy (CBT) protocols for procrastination with a wait-list control group. The interventions will be delivered online in group settings. Both protocols include identical psychoeducation and cognitive modules aiming at identification and modification of dysfunctional automatic thoughts related to procrastination but will differ in the behavioral modules. The behavioral module in the first protocol is focused on timely beginning and realistic planning. The second protocol implements working time restriction. The wait-list control group will receive one of the CBT protocols after a waiting period that will last as long as the CBT intervention and the assessments performed directly after treatment. It is assumed that the interventions will be superior to the wait-list control. Primary (procrastination) and secondary (depression and anxiety) measures will be collected prior to and after the interventions (or waiting period in the wait-list group) and after 6 months in the two active condition groups. Additionally, neuroimaging measurements will be conducted before and after the interventions (or waiting period in the wait-list group). Approximately half of the participants will undergo functional Magnetic Resonance Imaging (fMRI), and another half will undergo electroencephalography (EEG). Both methods are aimed at exploring neural correlates of the expected improvements in participants' self-regulation abilities.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor's and Master's university students
* Self-reported primary difficulties related to chronic and severe procrastination
* Serious procrastination problem lasting for at least one year as confirmed during clinical interview
* Having a postponed/procrastinated project to complete in the course of therapy
* Willing to participate in the study
* Fluent in Polish language
* Computer access and stable Internet connection

Exclusion Criteria:

* Current participation in other psychotherapy
* Use of psychiatric medication during the last 12 weeks
* Severe anxiety or affective disorders or any other severe psychiatric disorders that require other types of specialized care and are primary to procrastination problem (e.g. major depressive episode, social phobia, PTSD, etc.)
* Active suicidality
* Psychosis, bipolar disorder
* Alcohol or substance dependence
* Severe personality disorders (with the exclusion of avoidant, dependent and obsessive-compulsive personality disorders)
* For Warsaw participants: contradictions for fMRI measurement (metal elements in the body, claustrophobia, neurological conditions, pregnancy etc), non right-handedness.
* For Poznań participants: neurological conditions (e.g. epilepsy)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Polish version of the Pure Procrastination Scale (PPS) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of procrastination level. The Polish version of PPS consists of 12 items that evaluate procrastination conceptualized as a dysfunctional delay (e.g. "I am continually saying I'll do it tomorrow"; "I delay making decisions until it's too late"). Participants respond on a 5-point scale (1 = "very seldom or not true of me"; 2 = "seldom true of me"; 3 = "sometimes true of me"; 4 = "often true of me"; 5 = "very often true of true of me")
Change in Polish version of the Aitken Procrastination Inventory (API) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of academic procrastination level. The Polish version of API consists of 19 items that evaluate the tendency of students to procrastinate in their academic tasks (e.g. "If I had an important project to do, I'd get started on it as quickly as possible", "Getting down to work often takes me a long time."). Participants respond on a 5-point scale (1 = "false"; 2 = "mostly false"; 3 = " sometimes false/sometimes true"; 4 = "mostly true"; 5 = "true").

SECONDARY OUTCOMES:
Change in Polish version of the Patient Health Questionnaire (PHQ-9) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of depressive symptoms. The Polish version of PHQ-9 consists of 9 items that evaluate the occurrence of depressive symptoms in the last 2 weeks (e.g. "Little interest or enjoyment of your activities"). Participants respond on a 4-point Likert scale (0 = "not at all"; 1 = "on a few days"; 2 = "on more than half of the days"; 3 = "nearly every day").
Change in Polish version of the Generalized Anxiety Disorder Questionnaire-7 (GAD-7) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of anxiety symptoms. The Polish version of GAD-7 consists of 7 items that evaluate the occurrence of anxiety and excessive worry symptoms in the last 2 weeks (e.g. "Feeling afraid as if something awful might happen"). Participants respond on a 4-point Likert scale (0 = "not at all"; 1 = "on a few days"; 2 = "on more than half of the days"; 3 = "nearly every day").
Percentage of completion of a particular project that the participant decided to work on during the training (e.g. a thesis, an essay, a report). | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6)
  Before and after therapy they will be asked to assess the percentage of the project that has been completed. The higher the difference between the two assessments the better the outcome.

OTHER OUTCOMES:
Change in Polish version of the Sensitivity to Punishment and Sensitivity to Reward Questionnaire - Short Form (SPSRQ-SF) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Multidimensional-Multiattributional Causality Scale (MMCS) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Performance Failure Appraisal Inventory (PFAI) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Difficulties in Emotion Regulation questionnaire (DERS) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Motivation Diagnostic Test (MDT) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Zimbardo Time Perspective Inventory | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Metacognitive Beliefs about Procrastination Questionnaire (MBPQ) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Impulsivity Scale (UPPS-P) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Self-control Scale (NAS-50) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Procrastination Diagnostic Criteria Questionnaires (PDCQ) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of Positive and Negative Affect Schedule (PANAS) in relation to a project that the participant decided to work on during the training (e.g. a thesis, an essay, a report) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6
Polish version of the Group Session Rating Scale (GSRS) | During the intervention: at the end of every psychotherapy session (weeks 1-5)
Several items concerning homework compliance (cf. Kazantzis et al., 2005). | after sessions 2-5 (weeks 3-6) and at follow-up (6 months after post-treatment assessment)
Polish version of the Credibility Expectancy Questionnaire (CEQ) | After the first session (week 1)
Polish version of the Negative Effects Questionnaire (NEQ) | Post-treatment (week 6)
Polish version of the Client Satisfaction Questionnaire (CSQ) | Post-treatment (week 6)
fMRI measurements | baseline assessment (week 0), post-treatment assessment (week 6)
  Participants from Warsaw, prior to and after the interventions will undergo fMRI measurements, consisting of resting state and two cognitive tasks. In the first task participants will read sentences representing three conditions: sentences related to academic duties, sentences presenting negative events or situations, and sentences presenting neutral events or situations. The second task will be a monetary go/no-go task in two conditions: neutral condition, where participants will get some amount of money for each task block, regardless of their performance, and punishment condition, where participants will be given some amount of money prior to each task block, and will lose a fraction of the money each time when they respond to NoGo signal, or when they don't respond to Go signal or respond to it too slow.
Electroencephalography (EEG) measurements | baseline assessment (week 0), post-treatment assessment (week 6)
  Participants from Poznań before and after the interventions will undergo electroencephalography (EEG) measurements, during two emo-cognitive tasks. In the first task, participants will passively view single words related to three conditions: academic procrastination, negative emotions, neutral words. The second task will be a classic go/no-go task. In the posttest, there will be an additional negative norm-referenced feedback condition, where participants will be informed that their current performance in the go/no-go task is lower than a certain percentage of people who were tested. The EEG examination will utilize the Event-Related Potential (ERP) technique to measure the brain's electrical activity in response to specific events (stimuli and responses). This study will particularly focus on attentional processing and monitoring components, such as the P300, and Error Related Negativity (ERN) and Error Positivity (Pe).

CONTACTS AND LOCATIONS:
Overall Officials: Marek Wypych, PhD, DSc, Principal Investigator — Nencki Institute of Experimental Biology, Polish Academy of Sciences; Jarosław Michałowski, Prof., Principal Investigator — SWPS University of Social Sciences and Humanities; Joachim Kowalski, PhD, Principal Investigator — Institute of Psychology, Polish Academy of Sciences
Locations (1):
- Nencki Institute of Experimental Biology, Polish Academy of Sciences, Warsaw, Poland